CLINICAL TRIAL: NCT02529488
Title: Investigation of AcrySof® IQ PanOptix™ Presbyopia-Correcting IOL Model TFNT00
Brief Title: Investigation of AcrySof® IQ PanOptix™ Presbyopia-Correcting Intraocular Lens (IOL) Model TFNT00
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILH297-P002
Record Dates: First submitted 2015-08-19; First posted 2015-08-20 (Estimated); Results first posted 2018-04-06 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-03

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- TFNT00 (Experimental): AcrySof® IQ PanOptix™ Presbyopia-Correcting IOL, bilateral implantation
  Interventions: Device: AcrySof® IQ PanOptix™ Presbyopia-Correcting IOL

INTERVENTIONS:
Device: AcrySof® IQ PanOptix™ Presbyopia-Correcting IOL — Multifocal IOL(near, intermediate, distance) implanted for long-term use over the lifetime of the cataract patient
  Other Names: Model TFNT00

SUMMARY:
The purpose of this study is to investigate visual outcomes and assess safety at 12 months (330-420 days) post bilateral implantation of the AcrySof® IQ PanOptix™ Presbyopia-Correcting IOL.

DETAILED DESCRIPTION:
This study will be conducted in regions where the test article is approved at the time of study start.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bilateral cataracts with planned cataract removal by phacoemulsification with a clear cornea incision;
* Able to comprehend and willing to sign informed consent and complete all required postoperative follow-up procedures;
* Clear intraocular media other than cataract in both eyes;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Clinically significant corneal abnormalities including corneal dystrophy, inflammation or edema;
* Ocular trauma, corneal transplant, retinal conditions, degenerative eye disorders, or color vision deficiencies;
* Glaucoma (uncontrolled or controlled with medication) or ocular hypertension;
* Pregnant or lactating;
* Expected to require ocular surgical or retinal laser treatment;
* Other protocol-specified exclusion criteria may apply.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2015-09-07 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2017-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr Clinical Manager, Cataract, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 17 study centers located in Australia (4), Chile (3), Germany (2), Italy (2), Spain (2), Belgium (1), Great Britain (1), France (1), and Netherlands (1).
Pre-assignment Details: Of the 167 enrolled, 16 subjects were exited as screen failures prior to being implanted. An additional 2 subjects satisfied the eligibility criteria for the study, but were also discontinued prior to being implanted. This reporting group includes all implanted subjects (149).
Period: Overall Study
Arm/Group | TFNT00
Started | 149
Completed | 145
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Population: This analysis population includes all implanted subjects.
Arm/Group | TFNT00
Number analyzed (Participants) | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (9.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92
  Male | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43
  Not Hispanic or Latino | 100
  Unknown or Not Reported | 6

OUTCOME MEASURES:

1. Primary Outcome: Mean Binocular Defocus Visual Acuity (VA)
Description: Defocus VA (an indicator of the expected range of vision with a presbyopia-correcting IOL) was tested binocularly (both eyes together) with the subject's best spectacle correction at a distance of 4 meters. Lenses of different spherical powers were placed in front of the eyes to produce varying levels of defocus. The VA at each spherical power was measured in logarithm of the minimum angle of resolution (logMAR), with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an Early Treatment Diabetic Retinopathy Study (ETDRS) chart. A lower numeric value represents better visual acuity. The defocus VA summaries are based on the number of subjects evaluable for Best-Case Analysis Set and have data available at the corresponding visit. No formal statistical hypothesis testing was planned.
Time Frame: Day 20-40 and Day 120-180 from second eye implantation
Population: This analysis population includes all eyes successfully implanted with the test article that had at least 1 postoperative visit, no previous surgery for correction of refractive errors, no preoperative ocular pathology or macular degeneration at any time, no pregnancy during the study, and no major protocol deviations (Best-Case Analysis Set).
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- TFNT00 Visit 3A: AcrySof® IQ PanOptix™ Presbyopia-Correcting IOL, bilateral implantation at Day 20-40 post second eye implantation
- TFNT00 Visit 4A: AcrySof® IQ PanOptix™ Presbyopia-Correcting IOL, bilateral implantation at Day 120-180 post second eye implantation
Arm/Group | TFNT00 Visit 3A | TFNT00 Visit 4A
Number analyzed (Participants) | 137 | 134
logMAR
  +2.00 Diopter (D) | 0.570 (0.1893) | 0.569 (0.1844)
  +1.50D | 0.404 (0.1610) | 0.388 (0.1679)
  +1.00D | 0.209 (0.1386) | 0.214 (0.1413)
  +0.50D | 0.069 (0.1438) | 0.058 (0.1205)
  0.00D | -0.030 (0.1155) | -0.037 (0.1069)
  -0.50D | 0.037 (0.1099) | 0.043 (0.1180)
  -1.00D | 0.101 (0.1141) | 0.100 (0.1099)
  -1.50D | 0.072 (0.1175) | 0.065 (0.1302)
  -2.00D | 0.052 (0.1270) | 0.044 (0.1316)
  -2.50D | 0.077 (0.1396) | 0.066 (0.1338)
  -3.00D | 0.148 (0.1417) | 0.130 (0.1377)
  -3.50D | 0.257 (0.1532) | 0.256 (0.1551)
  -4.00D | 0.387 (0.1624) | 0.384 (0.1530)
  -4.50D | 0.495 (0.1674) | 0.491 (0.1583)
  -5.00D | 0.621 (0.1597) | 0.617 (0.1548)

ADVERSE EVENTS:
Time Frame: Test article implantation through study completion, an average of 1 year.
Description: Adverse Events (AEs) were obtained through volunteered and elicited comments from subjects and through observations by the Investigator. This analysis population includes all eyes with attempted test article implantation (successful or aborted after contact with the eye) (Safety Analysis Set). "At Risk" population of systemic AEs is reported in units of subjects; all other AE populations are reported in units of eyes.
Groups:
- TFNT00 - 1st Eye: All eyes with attempted test article implantation (successful or aborted after contact with the eye) in the 1st implanted eye
- TFNT00 - 2nd Eye: All eyes with attempted test article implantation (successful or aborted after contact with the eye) in the 2nd implanted eye
- TFNT00 - Non-Study Eye: All eyes not implanted with a study lens
- TFNT00 - Systemic: All subjects with attempted test article implantation (successful or aborted after contact with the eye).
Arm/Group | TFNT00 - 1st Eye | TFNT00 - 2nd Eye | TFNT00 - Non-Study Eye | TFNT00 - Systemic
All-Cause Mortality (participants affected / at risk) | 0/149 | 0/148 | 0/1 | 3/149
Serious Adverse Events (participants affected / at risk) | 3/149 | 4/148 | 0/1 | 11/149
Other Adverse Events (participants affected / at risk) | 21/149 | 21/148 | 0/1 | 0/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TFNT00 - 1st Eye (N=149) | TFNT00 - 2nd Eye (N=148) | TFNT00 - Non-Study Eye (N=1) | TFNT00 - Systemic (N=149)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 2 | 2 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Device dislocation (General disorders) | 0 | 1 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Intraocular pressure increased (Investigations) | 1 | 0 | 0 | 0
Optic nerve cup/disc ratio increased (Investigations) | 1 | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1
Visual field defect (Nervous system disorders) | 1 | 1 | 0 | 0
Eye operation (Surgical and medical procedures) | 1 | 0 | 0 | 0
Intraocular lens extraction (Surgical and medical procedures) | 1 | 0 | 0 | 0
Intraocular lens repositioning (Surgical and medical procedures) | 0 | 1 | 0 | 0
Joint arthroplasty (Surgical and medical procedures) | 0 | 0 | 0 | 1
Retinopexy (Surgical and medical procedures) | 2 | 1 | 0 | 0
Vitrectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TFNT00 - 1st Eye (N=149) | TFNT00 - 2nd Eye (N=148) | TFNT00 - Non-Study Eye (N=1) | TFNT00 - Systemic (N=149)
Dry eye (Eye disorders) | 15 | 13 | 0 | 0
Posterior capsule opacification (Eye disorders) | 6 | 8 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.